CLINICAL TRIAL: NCT04422795
Title: The Evaluation of External Thermomechanical Stimulation for Pain Reduction in Patients Undergoing Nail Injection
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to reallocation of resources, this study could not be initiated
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-03021647
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Nail Diseases
Keywords: Nails; Thermomechanical stimulation; Intralesional injection
MeSH Terms: conditions — Nail Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- External thermomechanical device delivering stimuli (Experimental): The thermomechanical device is placed on the digit proximally to the injection site with the ice wings frozen and the vibration mechanism switched on.
  Interventions: Device: External thermomechanical device delivering cold and vibration stimuli
- External thermomechanical device without delivering stimuli (Placebo Comparator): The thermomechanical device is placed on the digit proximally to the injection site with the ice wings at room temperature (unfrozen) and the vibration mechanism switched off.
  Interventions: Device: External thermomechanical device without delivering cold and vibration stimuli
- Nail injection with ethyl chloride skin refrigerant spray (Active Comparator): Ethyl chloride skin refrigerant spray is applied to the area of injection immediately before needle insertion
  Interventions: Drug: Ethyl chloride skin refrigerant spray

INTERVENTIONS:
Device: External thermomechanical device delivering cold and vibration stimuli — the thermomechanical device will be placed on the digit 2 cm proximally to the injection site with the ice wings frozen and the vibration mechanism switched on, delivering vibration and cold stimuli to the area for 30 seconds before the intramatricial injection and until needle withdrawal
  Arms: External thermomechanical device delivering stimuli
Device: External thermomechanical device without delivering cold and vibration stimuli — the thermomechanical device will be placed on the digit 2 cm proximally to the injection site with the ice wings at unfrozen and the vibration mechanism switched off, for 30 seconds before the intramatricial injection and until needle withdrawal
  Arms: External thermomechanical device without delivering stimuli
Drug: Ethyl chloride skin refrigerant spray — Ethyl chloride skin refrigerant spray is applied to the area of injection for 3 seconds immediately before needle insertion
  Arms: Nail injection with ethyl chloride skin refrigerant spray

SUMMARY:
The purpose of this study is to assess the efficacy and safety of a thermomechanical device delivering vibration and cold stimuli in lowering pain during intramatricial nail injections

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older
* Must understand and voluntarily sign an informed consent form
* All patients undergoing intramatricial nail injections at the Weill Cornell Medicine (WCM) Department of Dermatology
* Willingness to participate in the study

Exclusion Criteria:

* Inability of the patient to provide written informed consent for any reason
* Failure to have nail injection performed
* Likely inability to comply with the study protocol or cooperate fully with the research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The level of pain and change in pain between each time point will be assessed using the Wong-Baker FACES scale with use of thermomechanical device delivering stimuli, without delivering stimuli, and with use of ethyl chloride skin refrigerant spray. | prior to treatment, immediately after the needle insertion, during infiltration and 5 seconds after needle extraction
  Pain will be self-reported, using the Wong-Baker FACES (0-10, with 0 representing absence of pain and 10 unbearable pain). Participants will be questioned about their level of pain in their nail prior to treatment, immediately after the needle insertion, during infiltration, and 5 seconds after needle extraction

SECONDARY OUTCOMES:
Number of participants with at least one adverse event | Patients will be followed for 3 days following their nail injection
  Adverse events will only include those that are determined to be related to the study device

CONTACTS AND LOCATIONS:
Overall Officials: Shari R Lipner, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No